CLINICAL TRIAL: NCT05458258
Title: Investigating The Prognostic Significance Of Malnutrition And Sarcopenia In Older Adults With Acute Myeloid Leukemia
Brief Title: Studying Malnutrition And Sarcopenia In Older Adults With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB22-0397
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; Leukemia, Myeloid
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults (age 60+) with Newly Diagnosed AML: This group will consist of participants age 60+ who will be assessed for malnutrition and sarcopenia. Participants in this group will undergo chemotherapy and/or receive cancer drugs (as part of standard care). Participants in this group will receive different assessments when they start induction therapy to measure their nutritional health and the severity of their sarcopenia.
  Interventions: Device: Bioelectrical Impedence Analysis Device; Other: 6 Minute Walk Test; Diagnostic Test: Computed Tomography Scans to Measure Skeletal Muscular Index; Diagnostic Test: Blood Test/Blood Draw; Other: Hand Grip Strength Test
- Healthy Control Group: Adults with AML (age 60+) in Good Health: This group will also consist of participants age 60+ who will be assessed for malnutrition and sarcopenia. Participants in this group will undergo induction therapy and/or receive cancer drugs to treat their AML (as part of standard care). Participants in this group will also receive different assessments when they start induction therapy to measure their nutritional health and the severity of their sarcopenia. Participants in this group will receive the same assessment as participants in the first study group -- the only difference is that participants in this group have been determined to be healthier than those in the first study group according to clinical assessments.
  Interventions: Device: Bioelectrical Impedence Analysis Device; Other: 6 Minute Walk Test; Diagnostic Test: Computed Tomography Scans to Measure Skeletal Muscular Index; Diagnostic Test: Blood Test/Blood Draw; Other: Hand Grip Strength Test

INTERVENTIONS:
Device: Bioelectrical Impedence Analysis Device — A device that helps measure body composition, in particular body fat and muscle mass based on based on the rate at which an electrical current travels through the body.
Other: 6 Minute Walk Test — Defined as the distance the participant is able to walk in 6 minutes. Participants will be instructed to perform laps from the 0- to 30 minutes mark and back again for a total of 6 min in an outpatient or inpatient setting on a flat, pre-defined course. Participants will be instructed that goal of the test is to walk as far as possible.
Diagnostic Test: Computed Tomography Scans to Measure Skeletal Muscular Index — Computed tomography scans (a type of x-ray) that will measure the skeletal muscular index (the ratio of the muscle in your arms and legs to your height).
Diagnostic Test: Blood Test/Blood Draw — Blood will be drawn through a need inserted into the participant's arm. This blood will be used to measure the participant's nutrition levels.
Other: Hand Grip Strength Test — Grip strength in both hands will be measured using an adjustable hydraulic grip strength dynamometer (a device that is gripped to measure hand strength). The best performance of three trials will be selected for each hand, with averages of the left and right hand used in analyses.

SUMMARY:
This study will explore how malnutrition (poor nutrition/diet) and sarcopenia (a condition that causes a loss of muscle and bone mass) affects study participants over the age of 60 with acute myeloid leukemia (AML) who will receive induction chemotherapy (chemotherapy given as the first treatment to help cancer go into remission) and/or cancer drugs as part of standard care for AML. By studying how these nutritional and skeletal factors, doctors leading this study hope to learn how malnutrition and sarcopenia may be able to predict certain outcomes --such as how long study participants with poor nutrition and muscle loss can live after chemotherapy- for older (age 60+) individuals with AML.

ELIGIBILITY:
Inclusion Criteria:

* Older Adult patients (greater than or equal to 60 years of age)
* New diagnosis of acute myeloid leukemia (AML)
* Receiving induction therapy (intensive or low intensity therapy)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Presence of a pacemaker or defibrillator.
* Participants who are pregnant at the time of enrollment.
* Anyone unable/unwilling to follow protocol requirements

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with acute myeloid leukemia over the age of 60 who plan to receive induction therapy and/or cancer drugs for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Mortality Rates Based on Incidence of Sarcopenia in All Study Participants | 60 days
  This study's primary endpoint aims to measure the association of sarcopenia in study participants with their treatment-related mortality rate (how long the participant can stay alive 60 days after study treatment/registration). The incidence of sarcopenia in study participants will be measured using computed tomography-defined skeletal muscular index , hand grip strength test, and a 6-minute walk test. Treatment related mortality will be defined as the percent of patients no longer alive at 60 days after study registration.

SECONDARY OUTCOMES:
The prognostic impact of malnutrition and sarcopenia on treatment-related mortality rates and overall survival in study participants with AML | 60 days
  After pre-induction assessment (including assessments for sarcopenia and malnutrition), subjects will be prospectively followed for treatment-related mortality and overall survival assessments. Overall survival will be measured from date participants start on study to either death or last follow-up in accordance with 2017 European Leukemia Net recommendations. Treatment-related mortality rates will be defined as the percent of patients no longer alive at 60 days after registration.
Incidence of Malnutrition Among Participants in Group 1 Compared to Incidence of Malnutrition in Healthy Control Group | 60 days
  The incidence of malnutrition in older adults (≥60 years) with newly diagnosed AML undergoing intensive induction chemotherapy compared to the incidence of malnutrition in participants in the healthy control group. Incidence of malnutrition in both groups will be as assessed by participant questionnaires (known as subjective global assessments), blood tests , and Standardized bioelectrical impedance (BI) phase angle ( a measurement of the participant's body mass using a medical device).
Incidence of Sarcopenia Among Participants in Group 1 Compared to Incidence of Sarcopenia in Healthy Control Group | 60 days
  Incidence of sarcopenia in both study groups will be assessed by will be assessed by using computed tomography-defined skeletal mass index at L1, hand grip strength, and a 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States